CLINICAL TRIAL: NCT00372164
Title: Evaluation of the Effectiveness of Implementation of American Society of Interventional Pain Physician Guidelines for Interventional Techniques: A Retrospective Evaluation
Brief Title: Retrospective Evaluation of ASIPP Guidelines Implementation
Status: Withdrawn | Type: Observational
Sponsor: Pain Management Center of Paducah (Other)
Other Study IDs: protocol 14
Record Dates: First submitted 2006-09-01; First posted 2006-09-06 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Guideline Implementation
Keywords: ASIPP; Guidelines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: American Society of Interventional Pain Physician Guidelines

SUMMARY:
To demonstrate clinically significant improvements in the patients treated following ASIPP guidelines compared to the patients who were treated prior to the establishment of ASIPP guidelines.

DETAILED DESCRIPTION:
We have performed one study in the past showing that the implementation of guidelines improved outcomes by reducing the number of procedures and also the cost. However,, no large scale study has been performed thus far.

ELIGIBILITY:
Inclusion Criteria:

Evaluate all patients undergoing the following interventional techniques during 1999 and 2000 compared to patients undergoing interventional techniques during 2004 and 2005

* Cervical facet joint nerve blocks
* Thoracic facet joint nerve blocks
* Lumbar facet joint nerve blocks
* Lumbar interlaminar epidural steroid injections
* Cervical interlaminar epidural steroid injections

Exclusion Criteria:

Non-availability of appropriate data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: current patients
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 1998-01; Study Completion 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Laxmaiah Manchikanti, MD, Principal Investigator — Ambulatory Surgery Center
Locations (1):
- Ambulatory Surgery Center, Paducah, Kentucky, United States